CLINICAL TRIAL: NCT00523874
Title: Recurrence of Acute Alcoholic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Other Study IDs: R00126
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2001-01

CONDITIONS: Recurrent Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Previously our retrospective study showed that almost half of the patients with acute alcoholic pancreatitis had a recurrent attack in the long-term, mild pancreatitis and young age being risk factors for recurrence. The aim of this prospective follow-up study was aimed to find out the risk factors in detail.

DETAILED DESCRIPTION:
Patients admitted to Tampere University Hospital for first acute alcoholic pancreatitis were included. The diagnostic criteria for acute pancreatitis were epigastric pain, serum amylase > 3 x upper normal range, elevated serum CRP and signs of acute pancreatitis in imaging. Other etiologies were excluded. Alcohol consumption and dependency were detected. Serum and fecal markers of the endocrine and exocrine function and secretin stimulated MRCP were studied. The patients were followed median 38 (25 - 61) months for the recurrences and had a follow up visit at two years to investigate trends in the alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients who survived their first acute alcoholic pancreatitis. The diagnostic criteria for acute pancreatitis were epigastric pain, serum amylase > 3 x upper normal range, elevated serum CRP and signs of acute pancreatitis in imaging. Other etiologies were excluded.
* High alcohol consumption was detected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-01; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isto Nordback, MD,dos, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland